CLINICAL TRIAL: NCT05817344
Title: New Beginnings Following Trauma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Participant recruitment
Sponsor: Jesse McCann (Other)
Responsible Party: Sponsor-Investigator, Jesse McCann, Doctoral Student, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 81761
Record Dates: First submitted 2023-03-06; First posted 2023-04-18 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Stress Disorders, Post-Traumatic; Opioid Use Disorder
Keywords: Posttraumatic Stress Disorder (PTSD); Opioid Use Disorder (OUD); Written Exposure Therapy; Harm Reduction; Integrated Treatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Opioid-Related Disorders; Harm Reduction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3-Week Baseline (Experimental): Participants in this arm are randomized to a 3-week baseline period with repeated weekly assessment after the initial intake. Following the 3-week baseline, participants receive 5 weekly sessions of Written Exposure Therapy - Integrated (WET-I) followed by a 4-week follow-up phase with repeated weekly assessments.
  Interventions: Behavioral: Written Exposure Therapy - Integrated
- 5-Week Baseline (Experimental): Participants in this arm are randomized to a 5-week baseline period with repeated weekly assessment after the initial intake. Following the 5-week baseline, participants receive 5 weekly sessions of Written Exposure Therapy - Integrated (WET-I) followed by a 4-week follow-up phase with repeated weekly assessments.
  Interventions: Behavioral: Written Exposure Therapy - Integrated

INTERVENTIONS:
Behavioral: Written Exposure Therapy - Integrated — A brief exposure-based psychotherapy for posttraumatic stress disorder integrated with harm reduction strategies for opioid use disorder

SUMMARY:
Posttraumatic stress disorder (PTSD) is associated with increased rates of prescription opioid misuse, high-risk opioid use, illicit use of substances, and overdose (Meshberg-Cohen et al., 2021) Some research has demonstrated that among individuals with opioid use disorder (OUD), 92% report exposure to a traumatic event (Mills et al., 2005). Approximately 41% of those with OUD have a lifetime history of PTSD and 33.2% of individuals with OUD meet current diagnostic criteria for PTSD, indicating very high rates of PTSD among people with co-occurring OUD (Mills et al., 2006, 2007). PTSD also prospectively increases risk for OUD after exposure to opioids (Hassan et al., 2017).

Medications for opioid use disorder (MOUD) are evidence-based pharmacological interventions for OUD (methadone, buprenorphine, naltrexone) to manage pain and withdrawal (Leshner & Mancher, 2019). Though effective, dropout from MOUD programs is high (Mokri et al., 2016; O'Connor et al., 2020). It is also common in substance use disorder (SUD) treatment settings not to treat PTSD (Norman & Hien, 2020), though concurrent PTSD and MOUD treatment is associated with higher continuation in MOUD programs compared to no PTSD treatment (Meshberg-Cohen et al., 2019; Schacht et al., 2017). Despite this, there is little data regarding efficacy or effectiveness of specific trauma-focused PTSD treatments among patients in MOUD programs.

Combined with effective cognitive-behavioral techniques for substance use disorder (SUD), evaluation of brief, trauma-focused interventions for PTSD has substantial potential to improve care for individuals with PTSD receiving MOUD. The present study will begin to address this need by evaluating the feasibility, acceptability, and initial efficacy of Written Exposure Therapy (WET) for PTSD integrated with harm reduction skills for managing SUD symptoms among a sample of patients receiving MOUD [Written Exposure Therapy-Integrated (WET-I)]. WET is a five-session treatment for PTSD requiring limited therapist training and minimal patient burden (Sloan & Marx, 2019). WET has shown comparable outcomes to gold-standard interventions for PTSD, with improved retention rates (Sloan et al., 2018). WET has marked potential within this population, especially given that many clinicians in SUD programs do not have specialized training in PTSD treatments (Killeen et al., 2015).

Using a multiple baseline single case experimental design (SCED), 6 participants with current PTSD and current or past OUD will be recruited from MOUD treatment programs to engage in 5 weekly sessions of WET-I. Participants will complete an intake assessment to establish PTSD and OUD diagnoses and will be randomized to a 3- or 5-week baseline assessment period. Weekly assessments of symptoms (i.e., PTSD, anxiety, depression), substance craving and use, quality of life, and compliance with MOUD treatment will be completed during the baseline, treatment, and one-month follow-up phase. During the treatment phase, participants will also complete weekly measures of therapeutic alliance and will provide feedback on treatment credibility and treatment satisfaction.

Aim 1: To examine feasibility and acceptability of WET-I among participants in MOUD treatment with co-occurring PTSD/OUD. Feasibility of WET-I will be demonstrated via treatment retention and completion. Acceptability of engaging in WET-I in tandem with MOUD treatment will be demonstrated via high patient credibility ratings of WET-I and high treatment satisfaction ratings.

Aim 2: To determine if WET-I can significantly reduce symptoms of PTSD, anxiety, and depression in participants with comorbid PTSD and OUD and to monitor changes in drug use behaviors and craving over the treatment period. Participants will report reliable clinical improvement in symptoms (PTSD, anxiety, depression) and quality of life during the treatment phase and post-assessment without corresponding increases in substance use behavior or craving, and these improvements will be maintained at follow-up.

DETAILED DESCRIPTION:
Individuals interested in participating in this study will complete a phone screening or online screening based on individual preference to determine if they are likely to be eligible and can be scheduled for a telehealth or in-person diagnostic intake to take place at the Stress Trauma and Recovery Research Collaborative (STARRC) within the UK Clinic for Emotional Health. All participants will be provided with details regarding the screening questions and will be required to provide verbal consent over the phone or review a cover letter consent form (similar to the phone screening) online before proceeding with the screening. Once scheduled for an intake, participants will be sent a link to complete the intake questionnaires online prior to the start of the intake appointment. A cover letter consent form is attached for these questionnaires, as they will be administered before the in-person intake session. During the intake session, the participant will first be given a written and verbal description of the study and informed consent. The consent form will be presented to the participant on a tablet through REDCap, or via HIPAA-Compliant Zoom if telehealth, in which they will be asked to provide a digital signature. If consent is provided, they will be provided a copy. The PI or designated staff will discuss the informed consent form with the participant volunteer. The consent process will take place in a quiet and private room in our office or via HIPAA-Compliant Zoom. Participants may take as much time as needed to make a decision about their trial participation and may take the document home if desired. The person obtaining consent will thoroughly explain each element of the document and outline the risks and benefits, alternative treatment(s), and requirements of the study. Participants will be informed that they can withdraw from the research at any time.

Procedures and consent forms will comply with the requirements of the UK-IRB and ORI's Best Practices for Remote Informed Consent. The experimenter will then complete a consent post-test with participants. If a participant screens out of the study due to a consent capacity issue, any data from that participant that may have been previously collected during the phone screening and/or online surveys will not be used for research purposes and will be destroyed. Participants will also agree to the study's intoxication policy before signing the consent form. Participant privacy will be maintained and questions regarding participation will be answered. No coercion or undue influence will be used in the consent process. No research-related procedures will be performed prior to obtaining informed consent. All signatures and dates will be obtained. A copy of the signed consent will be given to the participant. Signed electronic consents will be maintained and stored through REDCap and will be separated from participant data.

After completing and signing the consent form at the intake appointment, eligible participants will be required to sign a release of information from the research team granting the research team permission to contact their methadone or buprenorphine program to coordinate care for the participant. Any additional release of information required from individual methadone or buprenorphine treatment facilities will be obtained for each participant as needed.

Initial Screening

Upon referral to the study, participants will complete a brief phone or internet screening based on participant preference to determine eligibility for an intake appointment. Screening forms for individuals who are deemed ineligible for the study for reasons other than consent capacity issues will be retained for study records and future research purposes that may be developed in the lab or by lab collaborators for which data may be useful.

First Baseline and Intake

Likely eligible participants, determined by the initial screen, will be asked to complete a battery of self-report questionnaires, which will assess for presence of DSM-5 psychological disorders, symptoms of anxiety/depression, level of functioning (e.g., quality of life), measures of PTSD, substance use, and substance craving (also to be completed online via REDCap). This survey platform is designed specifically for collection of research data, and therefore meets the privacy standards imposed on health care records by the Health Insurance Portability and Accountability Act (HIPAA). Referral information for resources to manage symptom difficulty will also be provided in the cover letter for these questionnaires. Likely eligible participants will be invited to attend the intake in-person or via telehealth in the PI's research lab at the Clinic for Emotional Health. A study assessor (i.e., doctoral students in clinical psychology/post-doctoral scholar/PI/Co-Is) will review study procedures with potential participants and ask them to provide their informed consent. After informed consent is provided, an interview-based diagnostic assessment will be administered in order to confirm clinical inclusion/exclusion criteria and urine and breathalyzer substance use screenings will be completed (for in-person participants only). This assessment visit will be video and/or audio-recorded. Recording via audio and/or video will be required for participation. Those who do not meet criteria for PTSD and/or other eligibility criteria will be told at the end of the assessment that they will not be able to continue in the study and will be provided referrals in-person or over email or postal mail for other treatment options depending on participant preference. Participants who do not endorse required eligibility criteria or who do endorse ineligibility criteria during the intake will not be permitted to continue in the study.

Baseline Period

Eligible participants will then be randomized to either a three- or five-week baseline where they will complete weekly measures of PTSD symptoms, symptoms of anxiety/depression, quality of life, substance use, and substance craving, and questions to determine whether they are in compliance with requirements of their MOUD program.

Treatment Period

The same questionnaire battery and substance use screenings will be repeated each week during therapy sessions, along with additional post-session ratings about treatment credibility and therapeutic alliance as well as interviews of substance use and urine and breathalyzer substance use screenings (for in-person participants). Urine and breathalyzer tests are standard operating procedure for studies assessing substance use behaviors in addition to self-reports of substance use.

Offering biological data to support participant self-reports is consistent with common research practices and will bolster scientific rigor of data reported in published manuscripts. If participants are completing treatment remotely, they will not complete substance use urine/breathalyzer screenings, but will still complete interviews of substance use via HIPAA-Compliant Zoom. Participants will then begin their first of five WET-I sessions. In WET, patients are provided with psychoeducation about trauma and PTSD in their first session and given explicit instruction on writing about the details of their most distressing trauma throughout treatment for 30 minutes each session followed by 10 minutes of structured discussion regarding the writing process. At the end of this discussion, therapists will introduce harm reduction strategies that will include 20 minutes of discussion in which therapists and participants will work together to establish and track the participant's goals for maintaining recovery over the next 5 weeks, discuss how engagement in WET-I can impact or cause barriers to these goals as well as ways in which the therapist can assist them in reducing barriers and achieving their goals, and discuss skills for safe substance use as needed (e.g., minimizing mixing substances, testing substances for fentanyl, using substances with people equipped to administer naloxone). The first session will be approximately 80 minutes while the remaining four will be approximately 60 minutes in length. Following completion of the treatment, participants will be asked to provide satisfaction ratings and written qualitative feedback on their experience with the treatment they received at the end of their last treatment session.

In order to bolster participation in weekly assessments, participants will be compensated up to $50 for each of the weekly baseline questionnaire batteries/drug screenings. If all assessments are not completed, they will receive funds for the amount of baseline assessments that they did complete. Participants will also receive up to an additional $50 for completion of each of the weekly questionnaire batteries during the treatment portion of the study. Participants will complete the same questionnaire/screening battery for three additional weeks following their post-treatment assessment one week after ending treatment.

It is important to note that the therapeutic strategies involved in WET-I are all common, evidence-based cognitive-behavioral strategies that have been shown to be safe among substance using populations. The treatment involves written exposures as instructed by an established manual (Written Exposure Therapy for PTSD) and brief processing of the exposure with the therapist. Treatment sessions will be audio- and/or video-recorded; this will allow study staff to rate sessions for fidelity to the protocol and will be used for clinical supervision. Recording via audio and/or video will be required for participation.

All self-report questionnaires will be completed online via REDCap. Questionnaires will be completed on-site using a study iPad or participants will be sent a link via email to complete the survey batteries during their own time. Finally, although investigators anticipate that most patients will prefer to complete these measures electronically, investigators can provide paper and pencil versions of the questionnaires if requested.

Data collection will be accomplished via screening questions, diagnostic interview, and self-report questionnaires attached below.

Through these measures investigators will collect data regarding participants' experiences with psychological symptoms, life functioning, and treatment satisfaction. Participants completing the study via telehealth will be sent REDCap links that to access the secure questionnaires that are specific to them.

The measures will be administered according to the following schedule:

Baseline, Intake, and Follow-Up Assessments:

Participants completing the intake session remotely or in-person will complete all of the same measures/assessments, with the exception of urine and breathalyzer screenings, which will only be completed by in-person participants.

Demographics - Intake and First Baseline Assessment, DIAMOND self-report screener - First Baseline Assessment, DIAMOND interview - Intake, Treatment Services Tracking Form - Intake, Last Follow-up Assessment, CSSRS/SAFE-T - Intake, AUDIT - First Baseline Assessment, DUDIT - First Baseline Assessment, Q-LES-Q - Weekly, TLFB - Weekly, Substance Craving - Weekly, PCL-5 - Weekly, ODSIS - Weekly, OASIS - Weekly, MOUD Compliance - Weekly, Urine and Breathalyzer Screenings - Weekly for in-person clients only

Pre-Session and Post-Treatment Assessment (Weekly):

Q-LES-Q - Weekly, PCL-5 - Weekly, TLFB - Weekly, Substance Craving - Weekly, ODSIS - Weekly, OASIS - Weekly, MOUD Compliance - Weekly, Treatment Services Tracking Form - First Therapy Session, Last Therapy Session, Urine and Breathalyzer Screenings - Weekly for in-person clients only, AUDIT - Post-Treatment Assessment, DUDIT - Post-Treatment Assessment

Post-Session (Weekly):

HAQ - Patient and Therapist - Weekly, CEQ (post-1st treatment session only), Patient Satisfaction Form (final treatment session only)

Investigators plan to utilize a randomized multiple baseline design across participants (Barlow et al., 2009; Kazdin, 2011). This is a form of single-case experimental design that provides a time and cost-effective method of evaluating initial efficacy or effectiveness of an intervention while controlling for the passage of time and repeated assessment in small numbers of patients. Patients will be randomized to either a 3- or 5-week baseline assessment phase where weekly self-report measures will be completed prior to initiating the treatment phase of the study. Randomizing to varying baseline periods enables assessments of whether symptoms change (only or more rapidly) when the intervention is applied (i.e., each participant acts as their own control). This design allows for causal inferences and controls for many threats to internal validity. Consistent with established guidelines, quantitative data analysis will primarily be conducted via visual inspection of graphed data within- and between-subjects to evaluate the magnitude and rate of change across the baseline and treatment phases (Barlow et al., 2009; Kazdin, 2011). This will be supplemented by examining within-person mean difference effect sizes for each outcome using a d-statistic developed for single case designs and calculating the percentage of patients who evidence reliable change on symptom measures (Jacobson & Truax, 1991; Shadish et al., 2014).

ELIGIBILITY:
Inclusion Criteria:

* History of trauma meeting past-month diagnostic criteria for posttraumatic stress disorder (PTSD; meeting diagnostic status on the DIAMOND PTSD Module and score greater than or equal to 36 on the PCL-5) and current or past diagnostic criteria for opioid use disorder (OUD).
* Enrolled in a methadone or buprenorphine treatment program in the state of Kentucky.
* 18 years of age or older and fluent in English (including being able to read and write in English).
* Participants on psychotropic medications and medications for opioid use disorder (methadone or buprenorphine) will be included if they have been maintained on a stable dose for at least 4 weeks prior to beginning the study and are willing to maintain a stable dosage throughout the study period; this procedure allows for a broader range of participants and avoids having outcomes assessment confounded by the initiation of medication during treatment.
* Participants in this study will also be required to sign a release of medical information for their methadone or buprenorphine clinic so that study staff can coordinate care with their methadone or buprenorphine provider.
* Willing to refrain from additional trauma-focused psychological treatment for the duration of the study.

Exclusion Criteria:

* Individuals diagnosed with psychological conditions that may be better addressed by alternative treatments. These conditions may include any history of psychotic disorders or dissociative identity disorder, manic episodes endorsed in the past year, current anorexia nervosa, and high risk of suicide.
* Individuals who endorse factors for which the treatment being studied (WET-I) may be contraindicated. These factors may include having no or limited memory of the trauma that would prevent the individual from engaging in written exposures.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-22 (Actual)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 | Change in PCL-5 scores will be assessed up to 14 weeks with self-report checklist from 3 or 5 weeks prior to beginning treatment, compared to weekly during treatment, and compared weekly to 4 weeks after completing treatment
  Change in Posttraumatic Stress Disorder Severity

CONTACTS AND LOCATIONS:
Overall Officials: Christal Badour, PhD, Study Director — University of Kentucky; Jesse McCann, MS, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Clinic for Emotional Health (CEH), Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No